CLINICAL TRIAL: NCT00593112
Title: A Pilot Study of Proton Magnetic Spectroscopy in Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD) Before and After Treatment With Osmotic-controlled Release Oral Delivery System (OROS) Methylphenidate
Brief Title: Proton Magnetic Spectroscopy in Children and Adolescents With ADHD Before and After Treatment With OROS Methylphenidate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paul Hammerness, MD, Clinical Investigator, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2005-P-002180
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Results first posted 2011-05-05 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: ADHD
Keywords: HMRS Scanning; ADHD; Child; Adolescent; HMRS Scans
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OROS Methylphenidate (Experimental)
  Interventions: Drug: OROS methylphenidate
- Control (Other): Healthy Volunteer Control group
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: OROS methylphenidate — Concerta is given in capsule form with a minimum dose of 18 mg/day and a max of 126 mg/day. Subjects take Concerta once per day for 6 weeks.
  Other Names: Concerta
  Arms: OROS Methylphenidate
Other: No intervention — No intervention
  Arms: Control

SUMMARY:
This will be an open label study using daily does of up to 126mg/day of Concerta in the treatment of children and adolescents, ages 12-17, who meet DSM-IV criteria for ADHD. Specific hypotheses are as follows:

Hypothesis 1: Children and adolescents with ADHD will have significantly higher ACC and DLPFC Glutamate/myo-Inositol containing compounds (Glu/Ino) and Glutamate/creatine + phosphocreatine (Glu/Cr) than matched HCS.

Hypothesis 2: After six weeks of treatment, OROS methylphenidate will lower ACC and DLPFC Glu/Ino and Glu/Cr levels in children with ADHD who are methylphenidate responders.

DETAILED DESCRIPTION:
The primary objective of this study is to use 1H MRS to assess Glutamate (Glu), myo-Inositol (Ino), and creatine + phosphocreatine (Cr) levels in brain regions of interest in 20 children with ADHD between the ages of 12-17 years old, before and after a six-week open treatment trial with OROS methylphenidate. For comparison, 1H MRS will also be obtained from 20 controls matched by age and gender. We also will scan 20 children with ADHD between the ages of 12-17 years old that are currently enrolled in the protocol entitled "Prevention of Cigarette Smoking in ADHD Youth with Concerta" (2003-P-001313) and on a stable dose of Concerta. These 20 children will be scanned once while on medication and once while off medication

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 12-17 years of age.
2. ADHD subjects must meet study criteria for the "Prevention of Cigarette Smoking in ADHD Youth with CONCERTA Protocol"; #2003-P-001313.
3. Control subjects must not meet full DSM-IV criteria for Attention Deficit Hyperactivity Disorder, or any other current major psychiatric disorder.
4. Each subject and his/her authorized legal representative must understand the nature of this proposed study, and must sign informed consent and informed assent documents.
5. Subject and parent must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with study procedures.

Exclusion Criteria:

1. Clinically significant chronic medical condition including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
2. Organic brain disorders or mental retardation (I.Q. <75).
3. Contraindication to MRI including presence of metal or surgical devices (plates, implants, braces or other items).
4. Pregnancy; women of child bearing potential must be using a medically approved method of birth control. Women of child bearing potential will receive a urinary pregnancy test prior to each MR scanning session.
5. Severe phobia of being in small, enclosed spaces.
6. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild will not be eligible to participate in the treatment arm of the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2006-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hammerness, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://massgeneral.org/pediatricpsych/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- OROS Methylphenidate: OROS = Osmotic-controlled Release Oral delivery System
Period: Overall Study
Arm/Group | OROS Methylphenidate | Control
Started | 27 | 12
Completed | 17 | 12
Not Completed | 10 | 0
Not completed — Scan Anxiety | 3 | 0
Not completed — Abnormal Scan | 1 | 0
Not completed — Unreadable Scan | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OROS Methylphenidate | Control | Total
Number analyzed (Participants) | 27 | 12 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 12 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 18 | 7 | 25
Region of Enrollment [Number; unit: participants]
  United States | 27 | 12 | 39

OUTCOME MEASURES:

1. Primary Outcome: Proton Magnetic Resonance Spectroscopy (H MRS) Scan Results - Glutamate(Glu)/Myo-inositol-containing Compounds (Ino)
Description: Comparison of treated ADHD participants (6 weeks on Concerta) and Healthy Control Subjects (HCS)
  This measure is a ratio of Glutamate (excitatory neurotransmitter) to myo-inositol (cyclic sugar alcohol) containing compounds in the anterior cingulate.
Time Frame: after 6 weeks Concerta treatment
Population: Seven subjects who completed the protocol were not included due to a lack of baseline comparison.
Measure: Mean (Standard Deviation); unit: MRS Ratio
Arm/Group | OROS Methylphenidate | Control
Number analyzed (Participants) | 10 | 12
MRS Ratio | 1.50 (0.45) | 1.56 (0.34)

2. Primary Outcome: H MRS Scan Results - Glutamine (Gln)/Ino
Description: Comparison of treated ADHD participants (6 weeks on Concerta) and Healthy Control Subjects (HCS)
  This measure is a ratio of Glutamine (amino acid precursor to Glu) to myo-inositol (cyclic sugar alcohol) containing compounds in the anterior cingulate.
Time Frame: after 6 weeks Concerta treatment
Population: Seven subjects who completed the protocol were not included due to a lack of baseline comparison.
Measure: Mean (Standard Deviation); unit: MRS Ratios
Arm/Group | OROS Methylphenidate | Control
Number analyzed (Participants) | 10 | 12
MRS Ratios | 1.08 (0.43) | 1.02 (0.60)

3. Primary Outcome: H MRS Scan Results - Glutamate & Glutamine (Glx)/Ino
Description: Comparison of treated ADHD participants (6 weeks on Concerta) and Healthy Control Subjects (HCS)
  This measure is a ratio of Glutamate and it's precursor, Glutamine, to myo-inositol (cyclic sugar alcohol) containing compounds in the anterior cingulate.
Time Frame: after 6 weeks Concerta treatment
Population: Seven subjects who completed the protocol were not included due to a lack of baseline comparison.
Measure: Mean (Standard Deviation); unit: MRS Ratio
Arm/Group | OROS Methylphenidate | Control
Number analyzed (Participants) | 10 | 12
MRS Ratio | 2.58 (0.73) | 2.59 (0.87)

ADVERSE EVENTS:
Arm/Group | OROS Methylphenidate | Control
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/12
Other Adverse Events (participants affected / at risk) | 0/27 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No